CLINICAL TRIAL: NCT02233270
Title: Validation of the AbStats Belt and Acoustic Esophago-Gastro-Intestinal Surveillance (AEGIS) System for Analyzing Motility Abnormalities
Brief Title: Pilot of AbStats /AEGIS System for Detecting Motility Abnormalities
Acronym: AEGIS
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mark Pimentel, MD, Director, GI Motility Program, Cedars-Sinai Medical Center
Other Study IDs: 32500
Record Dates: First submitted 2014-08-20; First posted 2014-09-08 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
When compared to existing analyses: manometry, Smart Pill and lactulose breath testing, external Acoustic Esophago-Gastro-Intestinal Surveillance (AEGIS) may identify unique audible patterns characteristic of features of gastroinestinal (GI) motility, gastric and small bowel contractions and emptying and small intestinal bacterial overgrowth (SIBO). This research study is designed to test the capabilities of AbStats/AEGIS to identify and associate symptoms and traditional diagnostics with sound readings and correlate this data with treatment outcomes and successes in standard of care.

DETAILED DESCRIPTION:
In partnership with Dr. William Kaiser and the UCLA Wireless Health Institute, our research groups are developing and validating the diagnostic capabilities of device that conducts AEGIS. A belt (AbStats) fits externally around the abdomen and is embedded with acoustic sensors, similar to "electronic stethoscopes." The investigational software is designed to continuously, safely, and comfortably monitor acoustic signals emanating from the esophagus, stomach, and intestines, and stores the data in a HIPAA compliant hard drive. Through the study of associating these readings with current diagnostics and treatments we anticipate that the AEGIS device will eventually provide clinically interpretable information that is immediately actionable. In this study, the Abstats sensor will track signals in tandem with current techniques and standard of care treatments based on those diagnostics. AEGIS analysis could potentially refine, support, or even replace, existing costly and invasive techniques in the diagnosis of gastroparesis, intestinal psueodo-obstruction, colonic inertia, and disorders related to small intestinal bacterial overgrowth (SIBO).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Scheduled for a small bowel manometry, SmartPill, or lactulose hydrogen breath test in the Cedars-Sinai Motility Program

Exclusion Criteria:

* Body mass index that is incompatible with placement of the belt (typically BMI greater than 45)
* Abdominal wall condition that disallows topical coverage as deemed by treating physician (eg abdominal wound, advanced cellulitis, draining ostomy etc)
* Inability to consent
* Have cognitive inability to follow directions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Cedars-Sinai Motility Program who are already scheduled to undergo small bowel manometry, SmartPill, or Lactulose Hydrogen Breath Test.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Acoustic readings of the abdominal cavity and swallowing collected via the device during current standard of care small bowel manometry reading. | At the time that the standard of care diagnostic test is performed, an expected average of 6 hours
  Acoustic readings would be recorded concurrent with standard of care diagnostics.
  There is no study follow up. Any patient follow up would be solely clinical standard of care, independent of study data or findings.
Acoustic readings of the abdominal cavity and swallowing collected via the device during current standard of care SmartPill transit recording. | At the time the standard of care diagnostic test is performed, up to 5 days
  Acoustic readings would be recorded concurrent with standard of care diagnostics.
  There is no study follow up. Any patient follow up would be solely clinical standard of care, independent of study data or findings.
Acoustic readings of the abdominal cavity and swallowing collected via the device during standard of care breath testing. | At the time the standard of care diagnostic test is performed, up to 3 hours.
  Acoustic readings would be recorded concurrent with standard of care diagnostics.
  There is no study follow up. Any patient follow up would be solely clinical standard of care, independent of study data or findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pimentel, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States